CLINICAL TRIAL: NCT00583258
Title: A Randomized, Double-Blinded Placebo-Controlled Trial of Alfuzosin (Xatral)in the Management of Distal Ureteral Calculi
Brief Title: A Randomized Study of Whether Alfuzosin(Xatral) Helps in the Passage of Kidney Stones
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SMHXATRAL2007; ALFUS-L-00811
Record Dates: First submitted 2007-12-20; First posted 2007-12-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Kidney Stones
MeSH Terms: conditions — Kidney Calculi | interventions — alfuzosin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Alfuzosin (Xatral)
- B (Placebo Comparator)
  Interventions: Drug: Placebo Alfuzosin

INTERVENTIONS:
Drug: Alfuzosin (Xatral) — 10 mg PO once a day
  Arms: A
Drug: Placebo Alfuzosin — 10 mg PO once a day
  Arms: B

SUMMARY:
Patients who present for the first time to Emergency Room with renal colic due to a distal ureteral calculus (as diagnosed with spiral CT scan and KUB) will be randomized to receive Xatral 10mg po once a day or placebo once discharged from the ER. The purpose of this study is to assess if patients treated with Xatral will have a higher spontaneous passage rate of their ureteral stone than those treated with placebo.

ELIGIBILITY:
Inclusion Criteria:

* first presentation to ER with renal colic secondary to a distal ureteral stone diagnosed on spiral CT scan
* stone radiopaque on KUB, distal to the sacro-iliac joint
* patient suitable for discharge from ER
* patient willing to return for follow-up on a weekly basis for maximum 4 visits

Exclusion Criteria:

* more than one ureteral calculi
* radiolucent stones or cystine stones
* prior ipsilateral calculus or ureteral surgery
* congenital anomalies of the ureter
* patients presents with an absolute indication for intervention
* allergy or contraindication to NSAIDs (history of orthostatic hypotension, current systolic BP <90 mmHg)
* patient currently taking an alpha-blocker
* hepatic insufficiency
* pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be Cox proportional hazards survival analysis of stone passage over time | 4 weeks

SECONDARY OUTCOMES:
Secondary outcomes will be stone passage rates, pain scores, intervention rates, hospitalization rates and complication rates | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth A Pace, MD, FRCSC, Principal Investigator — Unity Health Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada